CLINICAL TRIAL: NCT03759795
Title: Ameliorating the Impact of Complications and Errors on Surgeons: Resilience Training for Surgeons.
Brief Title: Bournemouth University Resilience Training for Surgeons
Acronym: BURTS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bournemouth University (Other)
Collaborators: Royal Bournemouth and Christchurch Hospitals NHS Foundation Trust (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 1819/IRASSR/1
Record Dates: First submitted 2018-11-13; First posted 2018-11-30 (Actual); Last update posted 2022-03-02 (Actual); Status verified 2022-03

CONDITIONS: Effect of Training
Keywords: Resilience; Psychological flexibility; Acceptance and Commitment Training

STUDY DESIGN:
Masking Description: Randomised Controlled Trial. Wait-list control for half participants. Other half receive ACTr (acceptance and commitment training) intention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): Acceptance and Commitment Training (ACTr)
  Interventions: Behavioral: ACTr (Acceptance and Commitment Training)
- Wait-list control (No Intervention): No intervention during trial. Participants in this group will be offered the training once the study is complete.

INTERVENTIONS:
Behavioral: ACTr (Acceptance and Commitment Training) — The programme is based on Acceptance and Commitment Training (ACT), a contemporary, empirically supported approach to psychological well-being.
  Arms: Intervention Group

SUMMARY:
The challenges that characterise surgical practice may result in a myriad of stressors that impact upon the personal and professional lives of surgeons. This includes a high likelihood that surgeons will have to deal with adverse patient outcomes due to surgical complications and errors, sometime during their careers. Such stressors can have undesirable effects on the surgeon in terms of quality of life and psychological well-being (e.g. anxiety, feelings of regret), as well as lowered professional confidence and impaired perceptions of professional competence. Furthermore, there is evidence that these kinds of negative impacts can also lead to burnout and depression. As well as the detrimental effects on surgeons and those around them, this in turn may lead to more errors and poorer outcomes for patients. This study will examine the efficacy of an ACT based training intervention to enhance resilience and psychological flexibility.

DETAILED DESCRIPTION:
Research in a range of occupational settings has indicated that resilience plays an important role in ameliorating the impact of adverse events in high pressure environments. This project will use a randomised controlled trial research design to assess the efficacy of brief one-to-one Acceptance and Commitment Training (ACTr), designed to enhance surgeons' psychological resilience. According to the model ACTr is based on, psychopathology is primarily the consequence of psychological inflexibility i.e. inability to persist or change behaviour according to long-term values due to language and cognition skills, which has particular significance when an individual is confronted with stress or adversity.

The main aim of this research is to assess the efficacy of a brief one-to-one Acceptance and Commitment Training course. Researchers wish to ascertain whether such a course can increase surgeons' resilience by increasing psychological flexibility, valuing and self-compassion (all of which are expected to be positively impacted by this training). This research will fill a gap in the relevant research literature; namely that no research project as far as we are aware has evaluated ACTr as a means to enhance resilience in surgeons. In fact any research conducted on resilience training with a surgical population is rare.

ELIGIBILITY:
Inclusion Criteria:

Trainee surgeons and consultant surgeons

Exclusion Criteria:

None

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2018-02-14 (Actual); Primary Completion 2022-01-01 (Actual); Study Completion 2022-01-01 (Actual)

PRIMARY OUTCOMES:
Resilience - Brief Resilience Scale (BRS) | 20 weeks
  A self-report measure of psychological resilience. Higher values represent a better outcome.
General Health - General Health Questionnaire (GHQ-12). | 20 weeks
  A self reported measure of minor psychological symptomology in a non-clinical population.

SECONDARY OUTCOMES:
CBI (Copenhagen Burnout Inventory) | 20 weeks
  A self-report measure of vulnerability to burnout. Lower values represent a better outcome.
DASS21 (Depression Anxiety and Stress Scale) | 20 weeks
  A self-report measure of depression, stress and anxiety. Lower values represent a better outcome.
VLQ (Value Living Questionnaire) | 20 weeks
  A self-report measure of valuing. Higher values represent a better outcome.
WAAQ (Work related Acceptance and Action Questionnaire) | 20 weeks
  A self-report measure of work related psychological flexibility. Higher values represent a better outcome.
AAQII (Acceptance and Action Questionnaire) | 20 weeks
  A self-report measure of general psychological inflexibility. Lower values represent a better outcome.
SCS (Self Compassion Scale) | 20 weeks
  A self-report measure of self compassion. Higher values represent a better outcome.
SPS (Sense of Preparedness Scale) | 20 weeks
  A self-report measure of preparedness for potential future events. Higher values represent a better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Helen Bolderston, Principal Investigator — Bournemouth University
Locations (2):
- United Kingdom (2):
  - Royal Bournemouth and Christchurch Hospitals NHS Foundation Trust, Bournemouth
  - Poole Hopsital, Poole

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Finnes A, Ghaderi A, Dahl J, Nager A, Enebrink P. Randomized controlled trial of acceptance and commitment therapy and a workplace intervention for sickness absence due to mental disorders. J Occup Health Psychol. 2019 Feb;24(1):198-212. doi: 10.1037/ocp0000097. Epub 2017 Sep 28. PMID 28956942
- [Background] Flaxman PE, Bond FW. A randomised worksite comparison of acceptance and commitment therapy and stress inoculation training. Behav Res Ther. 2010 Aug;48(8):816-20. doi: 10.1016/j.brat.2010.05.004. Epub 2010 May 8. PMID 20627269
- [Background] Pinto A, Faiz O, Davis R, Almoudaris A, Vincent C. Surgical complications and their impact on patients' psychosocial well-being: a systematic review and meta-analysis. BMJ Open. 2016 Feb 16;6(2):e007224. doi: 10.1136/bmjopen-2014-007224. PMID 26883234
- [Background] Shanafelt TD, Balch CM, Bechamps G, Russell T, Dyrbye L, Satele D, Collicott P, Novotny PJ, Sloan J, Freischlag J. Burnout and medical errors among American surgeons. Ann Surg. 2010 Jun;251(6):995-1000. doi: 10.1097/SLA.0b013e3181bfdab3. PMID 19934755
- [Background] Balch CM, Shanafelt TD, Dyrbye L, Sloan JA, Russell TR, Bechamps GJ, Freischlag JA. Surgeon distress as calibrated by hours worked and nights on call. J Am Coll Surg. 2010 Nov;211(5):609-19. doi: 10.1016/j.jamcollsurg.2010.06.393. Epub 2010 Sep 20. PMID 20851643
- [Background] Flaxman P. , Bond, F., Livheim, F. (2013): The Mindful and Effective Employee: An Acceptance and Commitment Therapy Training Manual for Improving Well-Being and Performance. New Harbinger Publications; 2013
- [Background] Turner, K., Johnson, C., Thomas, K., Bolderston, H., & McDougall, S. (2016). The impact of complications and errors on surgeons. The Bulletin Of The Royal College Of Surgeons Of England, 98(9), 404-407. doi: 10.1308/rcsbull.2016.404
- [Derived] Greville-Harris M, Wezyk A, Thomas K, Richer S, Bolderston H, Purchase N, McDougall S, Turner KJ. Acceptance and commitment therapy- based intervention to improve psychological skills and resilience in surgical trainees: a randomised waitlist-controlled trial. BMC Surg. 2025 Jul 28;25(1):315. doi: 10.1186/s12893-025-03059-5. PMID 40721794
- [Derived] Kunzler AM, Helmreich I, Chmitorz A, Konig J, Binder H, Wessa M, Lieb K. Psychological interventions to foster resilience in healthcare professionals. Cochrane Database Syst Rev. 2020 Jul 5;7(7):CD012527. doi: 10.1002/14651858.CD012527.pub2. PMID 32627860

DOCUMENTS (2):
  • Study Protocol (2018-06-11): https://cdn.clinicaltrials.gov/large-docs/95/NCT03759795/Prot_001.pdf
  • Informed Consent Form (2018-01-15): https://cdn.clinicaltrials.gov/large-docs/95/NCT03759795/ICF_000.pdf